CLINICAL TRIAL: NCT05534165
Title: Placebo-controlled Randomized Trial of Tecovirimat in Non-hospitalized Patients With Monkeypox: Canadian Feasibility Study (PLATINUM-CAN)
Brief Title: Tecovirimat in Non-hospitalized Patients With Monkeypox
Acronym: PLATINUM-CAN
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: The recommendations of the Data Safety Monitoring Committee, based on the results of the STOMP Study (NCT05534984).
Sponsor: Marina Klein (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); University Health Network, Toronto (Other); Unity Health Toronto (Other); University of British Columbia (Other); CIHR Canadian HIV Trials Network (Network)
Responsible Party: Sponsor-Investigator, Marina Klein, Professor of Medicine McGill University Health Centre, Research Director, MI4 Clinical Research Platform and Chronic Viral Illness Service, National Co-Director, CIHR Canadian HIV Trials Network, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTN 338
Record Dates: First submitted 2022-09-02; First posted 2022-09-09 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Monkeypox
Keywords: Tecovirimat; Randomized; Placebo-Controlled; Outpatients; Non-hospitalized; Feasibility
MeSH Terms: conditions — Mpox, Monkeypox | interventions — tecovirimat

STUDY DESIGN:
Intervention Model Description: Randomized 1:1
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Identical placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tecovirimat (Experimental): Tecovirimat (TPOXX®) Capsules, 200 mg (as tecovirimat monohydrate) administered as 600 mg (three 200 mg capsules) taken twice daily orally, every 12 hours, within 30 minutes after a full meal of moderate or high fat (approximately 25 g of fat) for 14 days
  Interventions: Drug: Tecovirimat
- Placebo (Placebo Comparator): Identical placebo supplied by SIGA Technologies Inc.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tecovirimat — 600 mg po BID
  Other Names: TPOXX
  Arms: Tecovirimat
Drug: Placebo — identical placebo 600 mg po BID
  Arms: Placebo

SUMMARY:
PLATINUM-CAN is a parallel collaborative trial linked with the sister trial PLATINUM led by Oxford University. PLATINUM-CAN is a multi-centre, randomized, placebo-controlled trial of Tecovirimat in non-hospitalized patients with presumptive or PCR confirmed monkeypox infection. The study will provide evidence on the efficacy and safety of Tecovirimat for laboratory-confirmed monkeypox in outpatients with monkeypox infection and determine the feasibility of conducting interventional monkeypox trials in Canada.

DETAILED DESCRIPTION:
In order to generate needed therapeutic efficacy evidence rapidly, international collaboration is essential. PLATINUM-CAN is a parallel collaborative trial linked with the sister trial PLATINUM led by Oxford University. Given the rapidly evolving epidemic and important differences in healthcare contexts and public health systems between countries that could impact the number of cases and access to diagnosis and treatment, a Canadian study is warranted to assess the feasibility and acceptability of conducting large scale interventional monkeypox trials in Canada. Such a focused trial also allows for the opportunity to explore a number of secondary objectives that can address concerns raised during consultation with Canadian community members (e.g., resolution of pain, quality of life) and validate use of self-assessed primary outcomes using blinded photography assessment.

The trial is pragmatic and minimizes number of visits, tests performed and contacts with the healthcare system through use of self-assessment diaries and self-testing. Lesion and/or throat swabs taken as part of standard care will be sent for detection of monkeypox virus DNA by PCR to local public health/provincial laboratories for initial screening (using panorthopox DNA testing) and confirmation with monkeypox specific PCR either locally or by National Microbiology Laboratory. The protocol allows for a broad range of patients to be enrolled. The trial has been designed so that it can accommodate patients who may be assessed in a variety of medical settings (e.g., hospital emergency rooms, outpatient HIV and infectious diseases clinics, community sexual health clinics, primary care, or through public health services). Similarly, we will ensure our trial design is able to contribute to global efforts such as the core protocol for the evaluation of treatments for human monkeypox (led by the Institut National de Recherche Biomédicale (INRB)/ANRS/NIAID in collaboration with WHO) and the AIDS Clinical Trials Group (ACTG) STOMP protocol.

As a feasibility study, PLATINUM CAN is underpowered for evaluating a primary endpoint of time to active lesion resolution. To achieve full study power, results will be combined with the sister study, PLATINUM-UK (n=500), being conducted at Oxford University, UK of similar design using a pre-planned individual patient meta-analysis. In addition to feasibility outcomes, the trial will evaluate the correlation between the time to active and complete resolution of lesions between self-report and blinded photographic validation from an adjudication committee, in consenting participants.

ELIGIBILITY:
Inclusion Criteria:

1. Any sex, ≥ 18 years of age inclusive at the time of signing informed consent.
2. Weight ≥ 40 kg
3. Laboratory-confirmed or presumptive monkeypox infection:

   Laboratory-confirmed monkeypox infection is defined as determined by PCR, culture, or antigen test obtained from a sample collected from blood, oropharynx, anal or skin lesion within 4 days of randomization OR

   Presumptive diagnosis:
   * Skin lesion(s), mucosal lesion(s) or proctitis consistent with a high probability of monkeypox infection in the opinion of the site investigator AND
   * Sexual contact with 1 or more persons in the 21 days prior to symptom onset or any person with known close exposure to another person known to be infected with monkeypox infection. Presence of active skin or mucosal lesion(s).
4. Appropriate to be managed without hospitalization.
5. The participant (or legally acceptable representative) has provided documented informed consent and comply to the require procedures for the study.

Exclusion Criteria:

1. Weight < 40 kg
2. Current or past use of tecovirimat
3. Inability to provide informed consent
4. The patient's own doctor considers there to be either a definite indication or a definite contraindication to the patient receiving tecovirimat
5. Participated in an interventional clinical study < 28 days prior to the day of first IP administration (Day 0) or plans to do so while enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Time to active lesion resolution | Up to 28 days after randomization
  Time (days) to active lesion resolution, defined as the first day on which all skin lesions are scabbed or desquamated (and mucosal lesions healed).
Feasibility and acceptability of conducting a pragmatic phase 3 interventional trial for outpatients with Monkeypox in Canada | 4 months
  Number of eligible patients per month and proportion randomized

SECONDARY OUTCOMES:
Time to complete lesion resolution | Up to 28 days after randomization
  Time (days) to complete lesion resolution, defined as the first day on which all lesions are completely resolved (all scabs dropped off and intact skin remains underneath, mucosal lesions healed)
Time to negative throat swab viral culture | Days 7, 14, 21, and 28
  Defined as time to consistently negative culture for monkeypox virus on throat swab
Time to negative skin or mucosa swab viral culture | Days 7, 14, 21, and 28
  Defined as time to consistently negative culture for monkeypox virus on swab of most recent active skin or mucosa
Secondary feasibility outcomes | 4 months
  the proportion who adhere to at least 85% of daily questionnaires and self-sampling, and the proportion of participants who are able to complete all protocol procedures

OTHER OUTCOMES:
Clinical status | day 7, 14, 21 and 28
  The ordinal scale is a) all lesions completely resolved (all scabs dropped off and intact skin remains underneath, mucosal lesions healed), b) all active lesions resolved (all lesions scabbed or desquamated, mucosal lesions healed), c) active lesions persist but no new lesions, d) new active lesions.
Throat swab monkeypox DNA levels | day 7, 14, 21 and 28
  Change from baseline in monkeypox virus DNA concentration in throat swabs
Hospitalization rates | study duration
  Number (%) of patients admitted to hospital for a complication of monkeypox, overall and by type
Time to sustained absence of use of analgesia | Up to 28 days post randomization
  defined as time to consistently reporting no use of analgesia
Assessment of safety | Duration of study
  1. Number (%) of patients suffering serious adverse events (overall and by type) up to 28 days of randomization
  2. Number (%) of patients suffering adverse events of special interest (overall and by type) up to 28 days of randomization
  3. Number (%) of patients suffering death, overall and by cause
Time to resolution of pain | 28 days
  Time to resolution of pain using an assessment for proctitis (rectal) and/or lesional pain comparing tecovirimat relative to placebo
Rate of improvement in overall quality of well-being | 28 days
  Change in EuroQol- 5 Dimension (EQ-5D) Quality Of Life scale
Validation of self reported time to active lesion resolution | 28 days
  Correlation between the time to active and complete resolution of lesions, in consenting participants, between self-report and blinded photographic validation from an adjudication committee

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - St. Paul's Hospital, BC Centre for Excellence in HIV/AIDS, Vancouver, British Columbia
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario